CLINICAL TRIAL: NCT02420795
Title: Phase I/II Study of Oral ONC201 in Patients With Relapsed/Refractory Non-Hodgkin's Lymphoma
Brief Title: Akt/ERK Inhibitor ONC201 in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per PI Request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0630; NCI-2015-00706 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 204666; 20152142; 1-909048-1; 1159132; 2014-0630 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2015-04-15; First posted 2015-04-20 (Estimated); Results first posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Central Nervous System Lymphoma; Gastric Mantle Cell Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma; Refractory Mantle Cell Lymphoma; Refractory Non-Hodgkin Lymphoma; Splenic Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Akt/ERK inhibitor ONC201) (Experimental): Patients receive Akt/ERK inhibitor ONC201 PO on day 1 of every cycle or day 1 of every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt/ERK Inhibitor ONC201; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt/ERK Inhibitor ONC201 — Given PO
  Other Names: ONC201; TIC10
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and the best dose of v-akt murine thymoma viral oncogene homolog (Akt)/mitogen-activated protein kinase 1(ERK) inhibitor ONC201 and to see how well it works in treating patients with non-Hodgkin's lymphoma that has returned after a period of improvement or does not respond to treatment. Akt/ERK inhibitor ONC201 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine recommended phase II dose for oral ONC201 (Akt/ERK inhibitor ONC201) in patients with relapsed/refractory lymphomas. (Phase I) II. To identify toxicities associated with oral ONC201 in patients with relapsed/refractory lymphomas. (Phase I) III. To determine the objective response rate to ONC201 in patients with relapsed/refractory lymphomas. (Phase II)

SECONDARY OBJECTIVES:

I. To determine the pharmacokinetics (PK) of oral ONC201 following administration. (Phase I) II. To observe the anti-tumor effects of oral ONC201, if any occur, in patients with relapsed/refractory lymphomas. (Phase I) III. Confirm tolerability of recommended phase II dose. (Phase II) IV. Assess clinical outcomes associated with ONC201 treatment in patients with relapsed/refractory lymphomas. (Phase II) V. Correlate clinical outcome with tumor and serum biomarkers. (Phase II)

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive Akt/ERK inhibitor ONC201 orally (PO) on day 1 of every cycle or day 1 of every week. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Phase 1 and Phase 2: confirmed diagnosis of previously treated relapsed and/or refractory lymphoma; patients with central nervous system (CNS) lymphoma are included
* Patient with leukemia phase (peripheral blood involvement), CNS lymphoma [including cerebrospinal fluid (CSF)-only disease], non-measurable disease, gastrointestinal (GI) mantle cell lymphoma (MCL), or bone marrow (BM) MCL are also eligible; gastrointestinal or bone marrow or spleen only patients are allowable and will be analyzed separately
* All adverse events related to prior therapies (chemotherapy, radiotherapy, and/or surgery) must be resolved to =< grade 1, except for alopecia
* Patients must be willing to receive transfusions of blood products
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or less
* Serum creatinine < 2.0 mg/dl
* Serum bilirubin < 1.5 mg/dl
* Platelet count > 50,000/mm^3
* Absolute neutrophil count (ANC) > 1,000/mm^3
* Alanine aminotransferase (ALT), or aspartate aminotransferase (AST) < 2 x upper limit of normal or < 5 x upper limit of normal if hepatic metastases are present
* Willing and able to participate in all study related procedures and therapy including swallowing capsules without difficulty
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test and must be willing to use acceptable methods of birth control during the study and for 90 days after the last dose of study treatment; acceptable methods of birth control include condoms with birth control foam, birth control pills, implantable or injectable birth control, birth control patch, intrauterine device (IUD), or diaphragm with spermicidal gel; male patients must use an effective barrier method of contraception (i.e. , condoms with birth control foam or diaphragm with spermicidal gel) during the study and for 90 days following the last dose of study treatment if sexually active with a female of childbearing potential; contraception must be in place at least 2 weeks prior to initiating study treatment; a female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must be English-speaking [MD Anderson Symptom Inventory (MDASI) completion only]

Exclusion Criteria:

* Any serious medical condition including but not limited to, uncontrolled hypertension, uncontrolled diabetes mellitus, uncontrolled infection, active/symptomatic coronary artery disease, chronic obstructive pulmonary disease (COPD), renal failure, active hemorrhage, or psychiatric illness that, in the investigators opinion places the patient at unacceptable risk or would prevent the subject from signing the informed consent form
* Pregnant or breast feeding females
* Use of any standard/experimental anti-lymphoma drug therapy, including steroids (dexamethasone dose >= 4 mg/day or prednisone >= 20 mg/day), within 3 weeks of initiation of the study or use of any experimental non-drug therapy (e.g., donor leukocyte/mononuclear cell infusions) within 56 days of initiation of the study drug treatment; hydroxyurea is permitted up to 24 hours before the first dose of study drug in patients with rapidly-proliferating disease
* Prior allogeneic stem cell transplant (SCT) within 16 weeks or autologous SCT within 8 weeks of initiation of therapy (patients that require immunosuppressive therapy are not eligible within 60 days of therapy)
* History of human immunodeficiency virus (HIV) infection; patients with active hepatitis B infection (not including patients with prior hepatitis B vaccination; or positive serum hepatitis B antibody); hepatitis C infection is allowed as long as there is no active disease and is cleared by GI consultation; HIV screening is not required for this study
* Significant neuropathy (grades 3-4, or grade 2 with pain) within 14 days prior to enrollment
* Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis, symptomatic inflammatory bowel disease, or partial or complete bowel obstruction, or any other gastrointestinal condition that could interfere with the absorption and metabolism of ONC201
* Major surgery within 4 weeks of initiation of therapy
* The patient has a prior or concurrent malignancy that in the opinion of the investigator, presents a greater risk to the patient's health and survival, than of the MCL, within the subsequent 6 months at the time of consent; investigator discretion is allowed
* Patients with New York Heart Association (NYHA) class III and IV heart failure, myocardial infarction in the preceding 6 months, and significant conduction abnormalities, including but not limited to second (2nd) degree atrioventricular (AV) block type II, third (3rd) degree block, QT prolongation (corrected QT [QTc] > 500 msec), sick sinus syndrome, ventricular tachycardia, symptomatic bradycardia (heart rate < 50 beats per minute [bpm]), hypotension, light headedness and syncope; patients with active atrial fibrillation will be excluded; the protocol excludes patients who have within the past year had a stent and by recommendation of their cardiologist need to stay on anticoagulants such as warfarin equivalent vitamin K antagonist
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ONC201 or its excipients
* Acute infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to initiation of study
* Active alcoholism or use of recreational drug (evaluated by history taking)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luhua (Michael) Wang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited at MD Anderson Lymphoma clinic from November 2015 through April 2018
Pre-assignment Details: A total of 16 participants consented for the protocol, 11 participated on the study, 4 of the participants were screen failures and 1 withdrew consent.
Groups:
- ONC201 125 mg: Patients receive Akt/ERK inhibitor ONC201 125 mg PO on day 1 of every cycle. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- ONC201 250 mg: Patients receive Akt/ERK inhibitor ONC201 250 mg PO every 7 days. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
- ONC201 625 mg: Patients receive Akt/ERK inhibitor ONC201 625 mg PO every 7 days. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | ONC201 125 mg | ONC201 250 mg | ONC201 625 mg
Started | 4 | 2 | 5
Completed | 0 | 0 | 0
Not Completed | 4 | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Progressive disease | 2 | 2 | 4
Not completed — Death | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Patients enrolled on Arm A until Arm B approved in 2/9/2016 IRB amendment
Groups:
- Total: Total of all reporting groups
Arm/Group | ONC201 125 mg | ONC201 250 mg | ONC201 625 mg | Total
Number analyzed (Participants) | 4 | 2 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 3 | 2 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 2 | 3
  Male | 3 | 2 | 3 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 2 | 4 | 9
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 2 | 5 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) (Phase I)
Time Frame: 21 days
Measure: Number; unit: mg
Groups:
- ONC201 125 mg: Patients receive Akt/ERK inhibitor ONC201 125 mg PO every 7 days. Cycles repeat every 21 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | ONC201 125 mg
Number analyzed (Participants) | 4
mg | 125

2. Primary Outcome: Number of Participants With Overall Response Rate (Phase 1 and 2)
Description: Defined as either progressive disease or stable disease observed assessed by the Revised International Workshop Standardization Response Criteria for non-Hodgkin lymphoma.
Time Frame: Up to 63 days (first 3 courses)
Population: 1 patient passed away prior to restaging in Phase 2 Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | ONC201 125 mg | ONC201 250 mg | ONC201 625 mg
Number analyzed (Participants) | 4 | 2 | 5
Participants
  Progressive Disease | 3 | 1 | 3
  Stable Disease | 1 | 1 | 1

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is the time in months from start of study treatment to date of death due to any cause.
Time Frame: every 3 months for 1 year, then every 6 months, up to 3 years
Population: Overall survival for each arm measured in months
Measure: Median (Full Range); unit: months
Arm/Group | ONC201 125 mg | ONC201 250 mg | ONC201 625 mg
Number analyzed (Participants) | 2 | 4 | 5
months | 29 [1 to 30] | 15 [1 to 30] | 24 [1 to 48]

4. Secondary Outcome: Progression-free Survival (PFS)- (Phase 2)
Description: Progression free survival is defined as time in weeks from start of study treatment to first documentation of objective tumor progression or up to death due to any cause, whichever occurs first.
Time Frame: every 3 months for 1 year, then every 6 months, up to 6 years
Measure: Median (Full Range); unit: weeks
Arm/Group | ONC201 625 mg
Number analyzed (Participants) | 5
weeks | 5 [1 to 10]

ADVERSE EVENTS:
Time Frame: From the first dose through every 3 months after the last dose of study medication, up to 1 year.
Arm/Group | ONC201 125 mg | ONC201 250 mg | ONC201 625 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 1/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/2 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ONC201 125 mg (N=4) | ONC201 250 mg (N=2) | ONC201 625 mg (N=5)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Dehydration (General disorders) | 0 | 1 | 0
Blood and lymphatic system disorders- Other (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial Infarction (Infections and infestations) | 0 | 0 | 1
Edema Limbs (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ONC201 125 mg (N=4) | ONC201 250 mg (N=2) | ONC201 625 mg (N=5)
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 1 | 0
Anxiety (Nervous system disorders) | 0 | 0 | 2
Appetite change (Metabolism and nutrition disorders) | 0 | 0 | 1
AST increased (General disorders) | 2 | 0 | 0
Back pain (General disorders) | 0 | 0 | 1
Blood and lymphatic system disorder (Blood and lymphatic system disorders) | 0 | 1 | 0
Blurred vision (Eye disorders) | 1 | 0 | 1
Bug bites (General disorders) | 0 | 0 | 1
BUN increased (Renal and urinary disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 4
Dizziness (Nervous system disorders) | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Ear Pain (Ear and labyrinth disorders) | 1 | 0 | 0
Edema limbs (General disorders) | 1 | 0 | 3
Edema trunk (General disorders) | 1 | 0 | 0
Elevated LDH (General disorders) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fatigue (General disorders) | 3 | 2 | 4
Fever (General disorders) | 0 | 0 | 1
GI bleeding (Gastrointestinal disorders) | 0 | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 0 | 1 | 0
Hematuria (Renal and urinary disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Memory changes (Psychiatric disorders) | 0 | 1 | 1
Memory impairment (Psychiatric disorders) | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2
Neutrophil count decreased (Investigations) | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Peripheral Sensory Neuoropathy (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 1 | 2
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Redness (both ears) (Eye disorders) | 1 | 0 | 0
Renal insufficiency (Renal and urinary disorders) | 1 | 1 | 0
Right carotid artery disease (General disorders) | 0 | 0 | 1
Runny nose (General disorders) | 0 | 1 | 0
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Splenomegaly (Infections and infestations) | 0 | 0 | 1
Thrush (Infections and infestations) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Weakness (General disorders) | 0 | 0 | 2
Weight loss (Investigations) | 0 | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Alkaline phosphatase increased (ALT) (General disorders) | 1 | 0 | 0
Left hip and thigh pain (General disorders) | 1 | 0 | 0
Left lower back pain (General disorders) | 1 | 0 | 0
Left lower leg pain (General disorders) | 1 | 0 | 0
Left quadrant abdominal pain (General disorders) | 1 | 0 | 0
Left shoulder pain (General disorders) | 1 | 0 | 0
Legs Muscle Cramps (General disorders) | 1 | 0 | 0
Loss of hearing on right ear (Ear and labyrinth disorders) | 1 | 0 | 0
Numbness (Nervous system disorders) | 1 | 0 | 0
Oral Thrush (Infections and infestations) | 1 | 0 | 0
Right Hip Pain (General disorders) | 2 | 0 | 0
Right Upper Quadrant Pain (General disorders) | 1 | 0 | 0
Numbness/Tingling (Nervous system disorders) | 0 | 2 | 0
Platelet Count Decreased (Blood and lymphatic system disorders) | 1 | 0 | 2
Acute abdominal pain on lower right (Gastrointestinal disorders) | 0 | 0 | 1
Chronic kidney disease (creatinine increased) (Renal and urinary disorders) | 0 | 0 | 1
Ecchymosis (bilateral forearms) (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Left ankle (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Sleep disturbance (Psychiatric disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/95/NCT02420795/Prot_SAP_000.pdf